CLINICAL TRIAL: NCT00000820
Title: A Phase II Study of Low-Dose Interleukin-2 by Subcutaneous Injection in Combination With Antiretroviral Therapy Versus Antiretroviral Therapy Alone in Patients With HIV-1 Infection and at Least 3 Months Stable Antiretroviral Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 248; 11225 (Registry Identifier: DAIDS ES Registry ID)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Interleukin-2; Drug Therapy, Combination; AIDS-Related Complex; Antiviral Agents
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — aldesleukin

INTERVENTIONS:
Drug: Aldesleukin

SUMMARY:
PRIMARY: To examine the effect of aldesleukin ( IL-2 ) on viral activity in the blood. To determine the safety of low-dose IL-2 in combination with antiretroviral therapy versus antiretroviral therapy alone.

SECONDARY: To examine delayed type hypersensitivity responses to skin test antigens and antibody responses to protein and polysaccharide vaccines.

The profound immune impairment that results from HIV-1 infection is due, at least in part, to the loss of CD4+ T cells and the cytokines these cells secrete, especially IL-2 and interferon-gamma. Antiretroviral agents do not directly address the problem of immune impairment. Replacement of IL-2 at nontoxic doses may prevent or delay clinical immunosuppression and its attendant opportunistic infections. Also, since patients with HIV-1 infection respond suboptimally to routine protein and polysaccharide immunizations, IL-2 may provide an adjuvant effect on vaccine responses.

DETAILED DESCRIPTION:
The profound immune impairment that results from HIV-1 infection is due, at least in part, to the loss of CD4+ T cells and the cytokines these cells secrete, especially IL-2 and interferon-gamma. Antiretroviral agents do not directly address the problem of immune impairment. Replacement of IL-2 at nontoxic doses may prevent or delay clinical immunosuppression and its attendant opportunistic infections. Also, since patients with HIV-1 infection respond suboptimally to routine protein and polysaccharide immunizations, IL-2 may provide an adjuvant effect on vaccine responses.

Patients are randomized initially to receive their own antiretroviral therapy alone or in combination with IL-2 for 24 weeks, after which each group is crossed over to the other treatment assignment (i.e., IL-2 is either added or deleted from the regimen) for an additional 24 weeks. Patients who are vaccine eligible receive influenza, tetanus and diphtheria toxoid, and meningococcal polysaccharide vaccines at week 4, and those who have not received pneumococcal vaccine prior to study entry will receive it at week 8.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* PCP prophylaxis.
* Therapy for an opportunistic infection that develops on study, with the exception of foscarnet for CMV disease or resistant Herpes simplex.
* Systemic corticosteroids ONLY IF given for no longer than 21 days for acute PCP.
* Topical corticosteroids to areas separate from a skin test or IL-2 injection site.
* Acyclovir up to 1000 mg/day as maintenance for recurrent genital Herpes.
* Erythropoietin and filgrastim.
* Antiemetics.
* Antibiotics as clinically indicated.
* Elective standard immunizations at week 8 or later.

Concurrent Treatment:

Allowed:

* Local radiation therapy.

Prior Medication: Required:

* Stable, approved antiretroviral therapy for at least 2 months (was 3 months, amended 3/26/96) prior to study entry.

Patients must have:

* HIV seropositivity.
* CD4 count 300 - 700 cells/mm3.
* Stable antiretroviral therapy for at least 2 months (was 3 months, amended 3/26/96) prior to study entry.
* No history of AIDS-defining illness except for limited cutaneous Kaposi's sarcoma.
* Normal EKG (isolated nonspecific ST and T wave changes permitted).

NOTE:

* This protocol is approved for prisoner participation.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Malignancy requiring systemic or local cytotoxic chemotherapy.
* Untreated thyroid disease.
* Asthma requiring intermittent or chronic inhalation or systemic therapy.
* Any medical condition that precludes study entry.

Concurrent Medication:

Excluded:

* Antianginal agents such as nitrates, calcium channel blockers, beta blockers, and antiarrhythmics.
* Systemic or local cytotoxic chemotherapy.
* Interferons.
* Interleukins other than study drug.
* Pentoxifylline ( Trental ).
* Acetylcysteine ( NAC ).
* Sargramostim ( GM-CSF ).
* Dinitrochlorobenzene ( DCNB ).
* Thymosin alpha 1.
* Thymopentin.
* Inosiplex ( Isoprinosine ).
* Polyribonucleoside ( Ampligen ).
* Ditiocarb sodium ( Imuthiol ).
* Therapeutic HIV vaccines.
* Investigational antiretroviral agents such as lamivudine ( 3TC ) and tat and protease inhibitors.
* Foscarnet.
* Aspirin.
* Immune globulin ( IVIG ).
* Thalidomide.
* Systemic corticosteroids (permitted for 21 days or less for PCP treatment only).

Concurrent Treatment:

Excluded:

* Ongoing transfusion.

Patients with the following prior conditions are excluded:

* History of autoimmune disease, including inflammatory bowel disease and psoriasis (although autoimmune thyroid disease that is stable is allowed).
* Clinically significant CNS disease or seizures that have been active within 1 year prior to study entry.

Prior Medication:

Excluded:

* IL-2 within 3 months prior to study entry.
* Any immunomodulatory therapy within 4 weeks prior to study entry.
* Foscarnet within 4 weeks prior to study entry.
* Acute therapy for an opportunistic infection within 14 days prior to study entry.

Active alcohol or substance abuse that would compromise study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104
Dates: Study Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teppler H, Study Chair; Pomerantz R, Study Chair
Locations (10):
- United States (10):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Cornell University A2201, New York, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Case CRS, Cleveland, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Vogler MA, Teppler H, Gelman R, Valentine F, Lederman MM, Pomerantz RJ, Pollard RB, Cherng DW, Gonzalez CJ, Squires KE, Frank I, Mildvan D, Mahon LF, Schock B; AIDS Clinical Trials Group 248 Study Team. Daily low-dose subcutaneous interleukin-2 added to single- or dual-nucleoside therapy in HIV infection does not protect against CD4+ T-cell decline or improve other indices of immune function: results of a randomized controlled clinical trial (ACTG 248). J Acquir Immune Defic Syndr. 2004 May 1;36(1):576-87. doi: 10.1097/00126334-200405010-00005. PMID 15097300